CLINICAL TRIAL: NCT06568445
Title: Efficacy of Regular ICS/LABA Sequential As-Needed Therapy in Newly Diagnosed Mild Asthma Patients: A Randomized, Parallel, Positive-Control Study
Brief Title: Maintenance at Initial Treatment With Sequential Anti-Inflammation Reliever Therapy
Acronym: MIT-AIR
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Zhou Yan, Deputy Chief Physician, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZYan
Record Dates: First submitted 2024-08-19; First posted 2024-08-23 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Bronchial Asthma
Keywords: asthma; budesonide-formoterol
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- maintenance at initial treatment sequential as-needed therapy group (Experimental): budesonide 160 µg-formoterol 4.5 µg (Symbicort 160/4.5) ®）, administered as one inhalation twice daily for maintenance for 4 weeks, sequential as-needed therapy for symptom relief to 24-week (no more than 8 inhalations per day).
  Interventions: Drug: Maintenance at initial treatment sequential as-needed therapy with inhaled budesonide-formoterol(Symbicort 160/4.5) ®）
- As-needed therapy group (Active Comparator): Inhaled budesonide-formoterol as needed when symptoms are present (Symbicort 160/4.5) ®），no more than 8 inhalations per day, continuous to 24-week.
  Interventions: Drug: as-needed therapy with inhaled budesonide-formoterol (Symbicort 160/4.5) ®）

INTERVENTIONS:
Drug: Maintenance at initial treatment sequential as-needed therapy with inhaled budesonide-formoterol(Symbicort 160/4.5) ®） — one inhalation twice daily for 4 weeks maintenance, sequential as-needed for symptom relief (no more than 8 inhalations per day) to 24-week.
  Other Names: maintenance at initial treatment sequential as-needed therapy group
  Arms: maintenance at initial treatment sequential as-needed therapy group
Drug: as-needed therapy with inhaled budesonide-formoterol (Symbicort 160/4.5) ®） — as-needed for symptom relief (no more than 8 inhalations per day) to 24-week.
  Other Names: As-needed therapy group
  Arms: As-needed therapy group

SUMMARY:
1. Evaluate the efficacy of 4 weeks of maintenance therapy with low-dose ICS/LABA versus as-needed low-dose ICS/LABA in newly diagnosed mild asthma patients. Assess the improvement in FEV1 from baseline over 4 weeks, and the impact on airway reversibility and inflammation levels. Identify the optimal patient population and treatment regimen for the medication.
2. Based on a comprehensive evaluation of pulmonary function parameters (including large airway parameters: FEV1, FEV1/FVC; peak flow: PEF; small airway parameters: FEF25%, FEF50%, FEF75%, MMEF) and airway inflammation levels, explore biomarkers that can effectively predict the efficacy of maintenance therapy with low-dose ICS/LABA in newly diagnosed mild asthma patients.
3. Compare 4 weeks of initial maintenance therapy with low-dose ICS/LABA followed by as-needed low-dose ICS/LABA therapy until 24 weeks. In the 24-week study, incorporate mobile lung function monitoring to dynamically assess large and small airway function parameters and clinical indicators. Explore the impact of early maintenance therapy with low-dose ICS/LABA followed by as-needed treatment on FEV1 improvement from baseline, acute exacerbation risk indicators, and airway inflammation, and develop a model to predict acute exacerbations.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients giving written informed consent will undergo a 1-week screening period to determine eligibility for study entry. At week 0, patients who meet the eligibility requirements will be randomized in a 1:1 ratio to research group (maintenance at initial treatment sequential as-needed therapy group) and control group (As-needed therapy group).

ELIGIBILITY:
Inclusion Criteria:

1. Participants fully understand the purpose and methods of the study, voluntarily agree to participate, and sign an informed consent form before any study procedures begin.
2. Adults (including males and non-pregnant, non-lactating females) aged 18 to 70 years (inclusive), who are newly diagnosed with mild and non-acute bronchial asthma according to the latest Chinese guidelines for the prevention and treatment of bronchial asthma.
3. During the screening period, participants must meet at least one of the following criteria for reversible airflow obstruction: Positive bronchodilator test (increase in FEV1 ≥12% and an absolute increase in FEV1 ≥200 mL after inhaling a bronchodilator). Positive bronchial provocation test (FEV1 decreases by ≥20% after inhalation of the provocation agent methacholine).
4. At screening and the Day -1 visit before the induction period, participants must have a lung function test showing FEV1 ≥ 80% of the predicted value.
5. Participants or their guardians must be able to communicate effectively with the researchers, understand, and comply with all requirements of the study.

Exclusion Criteria:

1. Individuals allergic or intolerant to budesonide, formoterol, albuterol, or any component of the medication.
2. Respiratory, sinus, or middle ear infections within the 2 months prior to screening or up to randomization that led to a change in asthma treatment, or are expected to alter the participant's asthma status according to the investigator's judgment.
3. History of chronic obstructive pulmonary disease (COPD), interstitial lung disease, restrictive lung disease, tuberculosis, cystic fibrosis, bronchiectasis, or alpha-1 antitrypsin deficiency at screening.
4. History of major diseases at screening, such as congestive heart failure, uncontrolled hypertension, severe coronary artery disease, myocardial infarction, or severe arrhythmias, or severe hematological, hepatic, neurological, musculoskeletal, endocrine, metabolic, psychiatric, renal, or other significant conditions. If any of these conditions worsen during the study, it may endanger the participant or affect study results.
5. Excessive use of short-acting beta-agonists (SABA), defined as more than 8 inhalations per day, during the screening period and the run-in period.
6. Use of beta-blockers (including eye drops), oral corticosteroids, systemic steroid treatments, investigational drugs, or leukotriene receptor antagonists (such as zafirlukast, pranlukast, montelukast, etc.) during the run-in period.
7. History of smoking with a smoking index >10 pack-years.
8. Smoking cessation ≤6 months before the screening visit (Visit 1) or current smokers.
9. Known or suspected alcohol and/or drug abuse, including heavy drinking (average daily consumption >2 units of alcohol, where 1 unit = 360 mL of beer, 45 mL of 40% alcohol, or 150 mL of wine).
10. Abnormal and clinically significant results in vital signs, physical examination, 12-lead ECG, chest CT, blood tests, urinalysis, blood biochemistry, or coagulation tests at screening and the Day -1 visit, unless judged by the investigator to be related to the study condition and not affecting inclusion.
11. Pregnant or breastfeeding females.
12. Use of medications that may interact with the study drug within 1 month before screening, such as CYP3A4 inhibitors (e.g., ketoconazole, itraconazole), cimetidine, disulfiram, metronidazole, or CYP3A4 enzyme inducers (e.g., rifampin, carbamazepine, phenytoin).
13. Participation in other medical device clinical trials within 1 month before screening or other drug clinical trials within 3 months before screening.
14. Asthma total symptom score (daytime + nighttime) <2 points in the week prior to randomization.
15. Patients who cannot comply with the study procedures or who, in the investigator's judgment, are not suitable for participation in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-08-12 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in forced expiratory volume in the first second (FEV1) at week 4 | Baseline and Week 4
  Spirometry was performed at baseline and after 4-week treatment, between 8:00 am and 10:30 am using MS-PFT spirometer (Jaeger, Hoechberg, Germany). Spirometry tests followed the standards of American Thoracic Society (ATS)/European Respiratory Society (ERS) recommendations. FEV1 is one pulmonary function parameter.

SECONDARY OUTCOMES:
Change from baseline in forced expiratory volume in the first second (FEV1) at Week 8, 12, 16, 20, 24 | Baseline and Week 8, 12, 16, 20, 24
  Spirometry was performed at baseline and after 8, 12,16, 20,24-week treatment, between 8:00 am and 10:30 am using MS-PFT spirometer (Jaeger, Hoechberg, Germany). Spirometry tests followed the standards of American Thoracic Society (ATS)/European Respiratory Society (ERS) recommendations. FEV1 is one pulmonary function parameter.
Change from baseline in Asthma control test (ACT) scrore | Baseline and Week 4, 8, 12, 16, 20, 24
  The ACT consists of 5 questions, each with a score ranging from 1 to 5 (for symptoms and activities: 1=all the time to 5= not at all; for asthma control rating: 1=not controlled at all to 5=completely controlled). The ACT score ranges from 5 (poor control of asthma) to 25 (complete control of asthma), with higher scores reflecting greater asthma control. ACT score ≥20 indicates well-controlled asthma.
Change from baseline in Asthma control questionnaire-5 (ACQ-5) | Baseline and Week 4, 8, 12, 16, 20, 24
  The ACQ-5 score was calculated as the mean score of 5 questions about asthma symptoms during the previous week. Each question is scored from 0 (no impairment) to 6 (maximum impairment), with higher scores reflecting poorer asthma control. ACQ-5 score >1.5 (asthma is poorly controlled), ACQ-5 score 0.75 -1.5 (asthma is partially controlled), ACQ-5 score <0.75 (asthma is well controlled).
Change from baseline in Fractional exhaled nitric oxide (FENO) | Baseline and Week 4, 8, 12, 16, 20, 24
  FENO was measured using NIOX MINO (Aerocrine AB, Solna, Sweden) at a standard flow rate of 50 ml/s following the ATS/ERS recommendations. FENO measurements were performed before spirometry and BCT since the involved breathing maneuvers may distort FENO results.
Change from baseline in Eosinophil counts in peripheral blood | Baseline and Week 4, 8, 12, 16, 20, 24
  Complete blood count (CBC) of peripheral blood was performed at baseline and after treatment by the clinical laboratory of Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine.
Change from baseline in Induced sputum classification and counting | Baseline and Week 4, 8, 12, 16, 20, 24
  Induced sputum method refers to inducing sputum production by inhaling nebulized hypertonic saline solution, and further analyzing the cellular components and soluble mediators in the supernatant of the sputum
Acute exacerbation of bronchial asthma | Week 4, 8, 12, 16, 20, 24
  Monitor the number of acute exacerbations of asthma, weeks of asthma symptom control, emergency medication, dosage of ICS and (oral corticosteroid) OCS, and use of background medication in patients after treatment.
Change from baseline in Forced Expiratory Flow at between 25% and 75% (FEF25%-75%) | Baseline and Week 4, 8, 12, 16, 20, 24
  FEF25%-75% is one pulmonary function parameter measured in spirometry.

OTHER OUTCOMES:
Adverse events | Week 4, 8, 12, 16, 20, 24
  Summarize the frequency, number, and incidence of the following adverse events by formulation group, severity, system organ classification (SOC), and preferred term for adverse events (PT): TEAE, TEAE related to the investigational drug. The incidence rate of adverse events shall be calculated at least once per subject for each SOC and PT.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Zhou, Principal Investigator — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai General Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
Sharing research plans, publishing data papers, and applying for patents

REFERENCES:
- [Background] Huang K, Yang T, Xu J, Yang L, Zhao J, Zhang X, Bai C, Kang J, Ran P, Shen H, Wen F, Chen Y, Sun T, Shan G, Lin Y, Xu G, Wu S, Wang C, Wang R, Shi Z, Xu Y, Ye X, Song Y, Wang Q, Zhou Y, Li W, Ding L, Wan C, Yao W, Guo Y, Xiao F, Lu Y, Peng X, Zhang B, Xiao D, Wang Z, Chen Z, Bu X, Zhang H, Zhang X, An L, Zhang S, Zhu J, Cao Z, Zhan Q, Yang Y, Liang L, Tong X, Dai H, Cao B, Wu T, Chung KF, He J, Wang C; China Pulmonary Health (CPH) Study Group. Prevalence, risk factors, and management of asthma in China: a national cross-sectional study. Lancet. 2019 Aug 3;394(10196):407-418. doi: 10.1016/S0140-6736(19)31147-X. Epub 2019 Jun 20. PMID 31230828
- [Background] Dusser D, Montani D, Chanez P, de Blic J, Delacourt C, Deschildre A, Devillier P, Didier A, Leroyer C, Marguet C, Martinat Y, Piquet J, Raherison C, Serrier P, Tillie-Leblond I, Tonnel AB, Tunon de Lara M, Humbert M. Mild asthma: an expert review on epidemiology, clinical characteristics and treatment recommendations. Allergy. 2007 Jun;62(6):591-604. doi: 10.1111/j.1398-9995.2007.01394.x. PMID 17508962
- [Background] Cloutier MM, Dixon AE, Krishnan JA, Lemanske RF Jr, Pace W, Schatz M. Managing Asthma in Adolescents and Adults: 2020 Asthma Guideline Update From the National Asthma Education and Prevention Program. JAMA. 2020 Dec 8;324(22):2301-2317. doi: 10.1001/jama.2020.21974. PMID 33270095
- [Background] Bergstrom SE, Boman G, Eriksson L, Formgren H, Foucard T, Horte LG, Janson C, Spetz-Nystrom U, Hedlin G. Asthma mortality among Swedish children and young adults, a 10-year study. Respir Med. 2008 Sep;102(9):1335-41. doi: 10.1016/j.rmed.2008.03.020. Epub 2008 Jul 17. PMID 18635346
- [Background] Crossingham I, Turner S, Ramakrishnan S, Fries A, Gowell M, Yasmin F, Richardson R, Webb P, O'Boyle E, Hinks TS. Combination fixed-dose beta agonist and steroid inhaler as required for adults or children with mild asthma. Cochrane Database Syst Rev. 2021 May 4;5(5):CD013518. doi: 10.1002/14651858.CD013518.pub2. PMID 33945639
- [Background] Beasley R, Holliday M, Reddel HK, Braithwaite I, Ebmeier S, Hancox RJ, Harrison T, Houghton C, Oldfield K, Papi A, Pavord ID, Williams M, Weatherall M; Novel START Study Team. Controlled Trial of Budesonide-Formoterol as Needed for Mild Asthma. N Engl J Med. 2019 May 23;380(21):2020-2030. doi: 10.1056/NEJMoa1901963. Epub 2019 May 19. PMID 31112386
- [Background] Hardy J, Baggott C, Fingleton J, Reddel HK, Hancox RJ, Harwood M, Corin A, Sparks J, Hall D, Sabbagh D, Mane S, Vohlidkova A, Martindale J, Williams M, Shirtcliffe P, Holliday M, Weatherall M, Beasley R; PRACTICAL study team. Budesonide-formoterol reliever therapy versus maintenance budesonide plus terbutaline reliever therapy in adults with mild to moderate asthma (PRACTICAL): a 52-week, open-label, multicentre, superiority, randomised controlled trial. Lancet. 2019 Sep 14;394(10202):919-928. doi: 10.1016/S0140-6736(19)31948-8. Epub 2019 Aug 23. PMID 31451207
- [Background] Busse WW, Pedersen S, Pauwels RA, Tan WC, Chen YZ, Lamm CJ, O'Byrne PM; START Investigators Group. The Inhaled Steroid Treatment As Regular Therapy in Early Asthma (START) study 5-year follow-up: effectiveness of early intervention with budesonide in mild persistent asthma. J Allergy Clin Immunol. 2008 May;121(5):1167-74. doi: 10.1016/j.jaci.2008.02.029. Epub 2008 Apr 11. PMID 18405951
- [Background] Selroos O, Pietinalho A, Lofroos AB, Riska H. Effect of early vs late intervention with inhaled corticosteroids in asthma. Chest. 1995 Nov;108(5):1228-34. doi: 10.1378/chest.108.5.1228. PMID 7587421
- [Background] Selroos O. Effect of disease duration on dose-response of inhaled budesonide in asthma. Respir Med. 2008 Jul;102(7):1065-72. doi: 10.1016/j.rmed.2007.12.029. Epub 2008 Apr 2. PMID 18387797
- [Background] O'Byrne PM, Pedersen S, Lamm CJ, Tan WC, Busse WW; START Investigators Group. Severe exacerbations and decline in lung function in asthma. Am J Respir Crit Care Med. 2009 Jan 1;179(1):19-24. doi: 10.1164/rccm.200807-1126OC. Epub 2008 Oct 31. PMID 18990678
- [Background] Henneberger PK, Patel JR, de Groene GJ, Beach J, Tarlo SM, Pal TM, Curti S. Workplace interventions for treatment of occupational asthma. Cochrane Database Syst Rev. 2019 Oct 8;10(10):CD006308. doi: 10.1002/14651858.CD006308.pub4. PMID 31593318
- [Background] Papi A, Canonica GW, Maestrelli P, Paggiaro P, Olivieri D, Pozzi E, Crimi N, Vignola AM, Morelli P, Nicolini G, Fabbri LM; BEST Study Group. Rescue use of beclomethasone and albuterol in a single inhaler for mild asthma. N Engl J Med. 2007 May 17;356(20):2040-52. doi: 10.1056/NEJMoa063861. PMID 17507703
- [Background] Martinez FD, Chinchilli VM, Morgan WJ, Boehmer SJ, Lemanske RF Jr, Mauger DT, Strunk RC, Szefler SJ, Zeiger RS, Bacharier LB, Bade E, Covar RA, Friedman NJ, Guilbert TW, Heidarian-Raissy H, Kelly HW, Malka-Rais J, Mellon MH, Sorkness CA, Taussig L. Use of beclomethasone dipropionate as rescue treatment for children with mild persistent asthma (TREXA): a randomised, double-blind, placebo-controlled trial. Lancet. 2011 Feb 19;377(9766):650-7. doi: 10.1016/S0140-6736(10)62145-9. Epub 2011 Feb 14. PMID 21324520
- [Background] Calhoun WJ, Ameredes BT, King TS, Icitovic N, Bleecker ER, Castro M, Cherniack RM, Chinchilli VM, Craig T, Denlinger L, DiMango EA, Engle LL, Fahy JV, Grant JA, Israel E, Jarjour N, Kazani SD, Kraft M, Kunselman SJ, Lazarus SC, Lemanske RF, Lugogo N, Martin RJ, Meyers DA, Moore WC, Pascual R, Peters SP, Ramsdell J, Sorkness CA, Sutherland ER, Szefler SJ, Wasserman SI, Walter MJ, Wechsler ME, Boushey HA; Asthma Clinical Research Network of the National Heart, Lung, and Blood Institute. Comparison of physician-, biomarker-, and symptom-based strategies for adjustment of inhaled corticosteroid therapy in adults with asthma: the BASALT randomized controlled trial. JAMA. 2012 Sep 12;308(10):987-97. doi: 10.1001/2012.jama.10893. PMID 22968888
- [Background] Sumino K, Bacharier LB, Taylor J, Chadwick-Mansker K, Curtis V, Nash A, Jackson-Triggs S, Moen J, Schechtman KB, Garbutt J, Castro M. A Pragmatic Trial of Symptom-Based Inhaled Corticosteroid Use in African-American Children with Mild Asthma. J Allergy Clin Immunol Pract. 2020 Jan;8(1):176-185.e2. doi: 10.1016/j.jaip.2019.06.030. Epub 2019 Jul 30. PMID 31371165
- See also: Related Info — http://www.ginasthma.org

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-06-25): https://cdn.clinicaltrials.gov/large-docs/45/NCT06568445/Prot_SAP_000.pdf
  • Informed Consent Form (2024-06-25): https://cdn.clinicaltrials.gov/large-docs/45/NCT06568445/ICF_001.pdf